CLINICAL TRIAL: NCT02938910
Title: Study of Myocardial Interstitial Fibrosis in Hyperaldosteronism Noninvasive Comparative Study in Humans of the Respective Cardiovascular Effects of Hyperaldosteronism and Hypertension by Magnetic Resonance Imaging
Brief Title: Study of Myocardial Interstitial Fibrosis in Hyperaldosteronism
Acronym: COEURALDO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110912
Record Dates: First submitted 2015-12-15; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Primary Hyperaldosteronism; Secondary Hyperaldosteronism; Essential Hypertension; Healthy
Keywords: Primary hyperaldosteronism; Secondary hyperaldosteronism; Cardiac fibrosis; magnetic resonance imaging
MeSH Terms: conditions — Hyperaldosteronism; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urines and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Volunteers: Healthy volunteers with normal blood pressure
  Interventions: Other: non interventional study
- Primary Hyperaldosteronism: Subjects with hypertension and high levels of seric aldosterone.
  Interventions: Other: non interventional study
- Secondary Hyperaldosteronism: Patient with Gitelman syndrome, with normal blood pressure and high level of aldosterone
  Interventions: Other: non interventional study
- Essential Hypertension: Patient with hypertension without secondary cause of hypertension
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study — Non invasive imaging study without interventional procedures

SUMMARY:
Animal models have demonstrated the role of aldosterone in left ventricular remodeling involving fibrosis, apoptosis and hypertrophy. Myocardial fibrosis is a risk factor for serious arrhythmia and sudden death in ischemic and idiopathic hypertrophic heart disease. It is accepted that patients with primary aldosteronism have a higher prevalence of LV hypertrophy , arterial involvement and increased cardiovascular risk. In humans, a link has been demonstrated between aldosterone and heart failure as well as the benefit of the administration of an anti -aldosterone drug to lower mortality in this population , regardless of blood pressure level . The administration of spironolactone ( aldosterone ) in hypertensive rats has prevented the occurrence of aortic fibrosis . Plasma aldosteronism in humans has been associated with inflammation, fibrosis and aortic stiffness . However, primary aldosteronism is generally associated with so-called secondary hypertension . Chronic hypertension alone is a recognized etiological factor of myocardial hypertrophy ( myocardial fibrosis very advanced ) . The purpose of this study is to investigate the effects of MRI hyperaldosteronism on the heart.

DETAILED DESCRIPTION:
Cross-sectional study with double analysis (A and B) with 2 x 2 sub-groups (ratio control/case 1/1)

* clinical situation: subjects are hypertensive. 20 subjects with primary aldosteronism will be compared to 20 patients with essential arterial hypertension
* clinical situation are normotensive subjects, 20 subjects with secondary aldosteronism loss in congenital salt (Bartter's syndrome / Gitelman) will be compared to 20 healthy volunteers. Controls (essential hypertension and healthy volunteers) are matched for age, sex and body size in two experimental groups (HAP and Gitelman). All subjects were recruited by the CIC of the European Georges Pompidou Hospital (Paris).

ELIGIBILITY:
* Patients with primary hyperaldosteronism:

  * Aldosterone / renin plasma ratio SUP 64 pmol / mU
  * aldosterone in a semi-sitting position SUP 500pmol / l or an aldosteronuria> 63nmol/24h,
  * Both under neutral treatment for at least 15 days (alpha-blocker, calcium channel blockers, central inhibitors). BMI = 35 kg / m².
* For patients with secondary hyperaldosteronism :

  * Documented diagnosis by the detection of mutation (s) homozygous or compound heterozygous for the gene SLC12A3 encoding CLCNKB chloride channel, or the gene encoding the HTSC Na-Cl cotransport thiazide sensitive.
  * Normal blood pressure (mean of three consecutive measurements of SBP INF 140 mmHg and DBP INF 90 mmHg measured in a semi-sitting position after 5 minutes of rest).
* For hypertensive patients :

  * Hypertension diagnosed on an average of three consecutive BP measurements = 140 and / or = 90 mmHg in the supine position after 5 minutes of rest or average daytime PA SUP 135/85 mmHg in ambulatory blood pressure monitoring (ABPM) in self-measurement , the presence of one or more antihypertensive medications regardless of the BP level.
  * No argument for secondary hypertension (renal artery stenosis, hypermineralocorticoidism, pheochromocytoma, iatrogenic ...) or negative balance of secondary hypertension.
  * BMI < 35 kg/m2.
* For healthy subjects :

  * Normal blood pressure (mean of three consecutive measurements of SBP INF 140 mmHg and DBP INF 90 mmHg measured in a semi-sitting position after 5 minutes of rest).
  * Absence of HA known or detected on determinations carried out during the study (see criteria for PAHs).
  * BMI <35 kg / m²
  * Laboratory tests (hematological and biochemical blood tests, urinalysis, serology and Research toxic) within normal limits or clinically acceptable for age and sex.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary hyperaldosteronism compared to hypertensive or normotensive controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Interstitial fibrosis assessed by MRI | One visit
  Quantitative interstitial fibrosis indices (intra- and extra-cellular LV mass) derived from myocardial relaxation time T1 MRI will be estimated in 4 populations with and without hypertension (patients with essential hypertension or with primary hyperaldosteronism versus healthy volunteers or patients with Gitelman syndrome), and with and without high level of aldosterone (patients with primary hyperaldosteronism or Gitelman syndrome versus patients with essential hypertension or healthy volunteers)

SECONDARY OUTCOMES:
Evaluation of myocardial remodeling by MRI | One visit
  Quantitative left ventricular remodeling (LV Mass and LV mass/end diastolic volume) will be estimated in 4 populations with and without hypertension (patients with essential hypertension or with primary hyperaldosteronism versus healthy volunteers or patients with Gitelman syndrome), and with and without high level of aldosterone (patients with primary hyperaldosteronism or Gitelman syndrome versus patients with essential hypertension or healthy volunteers)
Effect of hypertension on myocardial fibrosis assessed by MRI | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between the degree of myocardial fibrosis
Effect of aldosteronism on myocardial fibrosis assessed by MRI | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between the degree of myocardial fibrosis
Effect of hypertension on LV diastolic dysfunction | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between the degree of LV diastolic dysfunction
Effect of aldosteronism on LV diastolic dysfunction | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between the degree of LV diastolic dysfunction
Effect of hypertension on the relationship between circulating biomarkers of fibrosis | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between circulating biomarkers of fibrosis
Effect of aldosteronism on the relationship between circulating biomarkers of fibrosis | One visit
  Analyze the relationship in each of the two clinical situations (HTA or absence of hypertension) between circulating biomarkers of fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Elie MOUSSEAUX, MD, PhD, Study Director — Assistance publique des hopitaux de Paris; Alban REDHEUIL, MD,PhD, Study Director — Assistance publique des hopitaux de Paris
Locations (1):
- Centre d'investigation Clinique, hopital Europeen George Pompidou, Paris, France

REFERENCES:
- [Derived] Redheuil A, Blanchard A, Pereira H, Raissouni Z, Lorthioir A, Soulat G, Vargas-Poussou R, Amar L, Paul JL, Helley D, Azizi M, Kachenoura N, Mousseaux E. Aldosterone-Related Myocardial Extracellular Matrix Expansion in Hypertension in Humans: A Proof-of-Concept Study by Cardiac Magnetic Resonance. JACC Cardiovasc Imaging. 2020 Oct;13(10):2149-2159. doi: 10.1016/j.jcmg.2020.06.026. Epub 2020 Sep 16. PMID 32950448